CLINICAL TRIAL: NCT01763060
Title: Long Term Follow up of Patients Who Were Treated With Extracorporeal Membrane Oxygenation for Pandemic Influenza A/H1N1 Induced Severe Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Bernhard Holzgraefe, MD, Karolinska University Hospital
Other Study IDs: Dnr 2012/986-31/3; Long term outcome (Other: Ehtical committee Stockholm)
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Long Term Outcome
Keywords: ards; ecmo; h1n1; pandemics
MeSH Terms: conditions — Acute Lung Injury | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ECMO survivors: CT scan of the chest of all ECMO survivors after 2009/2010 pandemics Tests for cognitive function MRI of the brain Lung function
  Interventions: Radiation: CT scan; Behavioral: Cognitive function; Radiation: MRI

INTERVENTIONS:
Radiation: CT scan
Behavioral: Cognitive function
Radiation: MRI

SUMMARY:
Patients treated with Extracorporeal Membrane Oxygenation (ecmo) for severe respiratory or circulatory failure show severe long term disability due to impaired lung -, cerebral-, cognitive function and impaired quality of life. This study investigates the long term outcome of all patients who are still alive three years after ECMO treatment for severe respiratory failure during the H1N1 2009 pandemic at the Karolinska University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of ECMO treatment for influenza a/h1n1 pneumonia during 2009/2010 pandemics at the ECMO Center Karolinska

Exclusion Criteria:

* None

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: All patients who survived ECMO treatment due to infection with Influenza A/H1N1 2009 up to 3 years after discharge from hospital
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Lung function | 3 years after ecmo treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Holzgraefe B, Andersson C, Kalzen H, von Bahr V, Mosskin M, Larsson EM, Palmer K, Frenckner B, Larsson A. Does permissive hypoxaemia during extracorporeal membrane oxygenation cause long-term neurological impairment?: A study in patients with H1N1-induced severe respiratory failure. Eur J Anaesthesiol. 2017 Feb;34(2):98-103. doi: 10.1097/EJA.0000000000000544. PMID 28030441